CLINICAL TRIAL: NCT05179642
Title: Impact of a Consultation Between a Coordinating Physician and a Referring Physician About the Optimization of Drug Prescription for Each Resident Entering in Nursing Home (EHPAD).
Brief Title: OPTIM-EHPAD Optimization of Drug Prescription for Each Resident Entering in Nursing Home (EHPAD).
Acronym: OPTIM-EHPAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0009
Record Dates: First submitted 2021-11-08; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-11

CONDITIONS: Iatrogenic Effect
Keywords: coordinating physician; referring physician; optimization of drug prescription; nursing home; inappropriate prescription

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: This is a randomized, cluster stepped wedge study. The cluster will be made up of coordinating physicians grouped together according to the geographical area of their EHPAD.
  Residents entering EHPAD during the pre-interventional inclusion period will be treated as usual in EHPAD. They will constitute the control group.
- Tool OPTIM-EHPAD: This is a randomized, cluster stepped wedge study. The cluster will be made up of coordinating physicians grouped together according to the geographical area of their EHPAD.
  Residents entering EHPAD during the post-intervention inclusion period will have the optimization of their diagnostic and drug management, following a consultation between their referring physician and the coordinating physician based on the OPTIM-EHPAD method. They will constitute the intervention group.
  The intervention is based on the utilization of the OPTIM-EHPAD method. It consists in training for coordinating physician and, optionally, for referring physician. It's a pedagogic tool proposing a rigorous methodology for reviewing prescriptions in chronological stages, associated with memos, constituting a form of clinical path for improving the quality and safety of prescriptions for EHPAD residents.
  Interventions: Other: OPTIM-EHPAD tool

INTERVENTIONS:
Other: OPTIM-EHPAD tool — This is a randomized, cluster stepped wedge study. Residents entering EHPAD during the pre-interventional inclusion period will be treated as usual in EHPAD. They will constitute the control group.
  Residents entering EHPAD during the post-intervention inclusion period will have the optimization of their diagnostic and drug management, following a consultation between their referring physician and the coordinating physician based on the OPTIM-EHPAD method. They will constitute the intervention group.
  The intervention is based on the utilization of the OPTIM-EHPAD method. It consists in training for coordinating physician and, optionally, for referring physician. It's a pedagogic tool proposing a rigorous methodology for reviewing prescriptions in chronological stages, associated with memos, constituting a form of clinical path for improving the quality and safety of prescriptions for EHPAD residents.
  Groups: Tool OPTIM-EHPAD

SUMMARY:
Elderly people are at high risk of multiple medication which increases drug interactions and side effects. This problem is accentuated in EHPAD due to the multiplication of prescribers (the referring physician, the hospital physician, the specialist, the emergency physician, the coordinating physician). The lack of optimization of drug prescriptions in EHPAD can be responsible for iatrogenic, underuse and overuse of treatment, impacting the autonomy and quality of life of residents in EHPAD in France.

A method for optimizing diagnostic and drug management at the entry of a new EHPAD resident, called OPTIM EHPAD, has been tested in Languedoc-Roussillon (France) and validated. This is a consultation between the referring physician and the EHPAD coordinating physician. Some improvements have been made to this method in order to have an optimized version.

Physician's cooperation seems to promote decision-making and change in therapies. The objective of this study is to assess the theoretical effectiveness and efficiency of this approach.

It is supposed that the provision to the EHPAD coordinating physician of a method for optimizing the diagnostic and drug management of the new EHPAD resident (based on a decision following consultation between the referring doctor and the coordinating doctor) would impact on the resident care process, on their care results and on communication and coordination between the coordinating physician and the referring physician.

ELIGIBILITY:
Inclusion Criteria:

* - Coordinating physician of EHPAD who don't have an indoor pharmacy (PUI) from the Languedoc-Roussillon-Midi-Pyrénées region and the Auvergne-Rhône-Alpes region.
* New resident entering a participating EHPAD

Exclusion Criteria:

* - Residents who don't have a referring physician when entering EHPAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible population is made up of EHPAD coordinating physicians who don't have an indoor pharmacy (PUI) from the Languedoc-Roussillon-Midi-Pyrénées region and the Auvergne-Rhône-Alpes region.
  Any new resident entering a participating EHPAD. Residents who don't have a referring physician when entering EHPAD will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Inappropriate prescription line and average number of days of hospitalization | 6 months after the entering patient in EHPAD
  hierarchical sequential approach on the following criteria according to the predefined order :
  1. Proportion of residents with at least one inappropriate prescription line in residents' drug dispensations during months M3 to M6 following their entry into EHPAD.
  2. Average number of days of hospitalization per resident in internal medicine/surgery/obstetrics wards, follow-up care and rehabilitation or in a psychiatric establishment during the 6 months following entry into EHPAD

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France